CLINICAL TRIAL: NCT07297680
Title: Workplace Exercises Versus Home-based Exercises on Pain and Function Among Office Workers With Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Allah Ahmed Gaber Abd El Tawab, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Heba-Msc
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain; Pain; Function; Office Worker; Workplace Exercise; Home Bases Exercise
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- workplace exercise (Experimental): Consists of 20 office workers with non-specific low back pain who will receive workplace exercise intervention, 5 times per week for 4 weeks
  Interventions: Other: Workplace exercise intervention
- home program exercises (Active Comparator): Home program exercises will be provided three times a week for four weeks, comprising three sets of ten repetitions each. Exercises will target the back, shoulders, and arms using elastic tubing, including reverse flys, shoulder raises, shoulder squeezes, shoulder rotations, wrist extensions, wood choppers, pelvic tilt, quadruped leg/arm raises, side planks, and lean and turns.
  Interventions: Other: Home-based exercise intervention
- general education and counseling (Active Comparator): Individuals will receive education and counseling on managing pain and function. They should avoid prolonged sitting, moving every 20-30 minutes, and practicing good posture while seated, standing, and walking. Key sitting posture includes keeping feet flat, knees at a 90-degree angle, and maintaining a straight back with proper lumbar support to prevent slouching.
  Interventions: Other: general education and counseling

INTERVENTIONS:
Other: Workplace exercise intervention — The program's basic exercise equipment includes a stable chair (no wheels or armrests) that provides better lumbar spine support, adjustable for participant height to ensure flat feet on the floor with a 90° knee angle. Additional portable equipment consists of a rhythmic gymnastics ball (16.5 cm diameter, 320 g weight), silicone hand therapy balls (5.6 cm length, 4.2 cm width, medium resistance), and an exercise band (1.5 m long, available in medium/light and heavy resistance).
  Arms: workplace exercise
Other: Home-based exercise intervention — An elastic exercise band will be used. an exercise band (1.5 m long, available in medium/light and heavy resistance).
  Arms: home program exercises
Other: general education and counseling — Will receive general education and counseling regarding pain and function. They will be advised to avoid prolonged sitting. Get up and move around every 20-30 minutes. In addition, to practice good posture while sitting, standing, and walking. When sitting, keep your feet flat on the floor, knees bent at a 90-degree angle, and your back straight with good lumbar support. Furthermore, to avoid slouching or hunching over their desk
  Arms: general education and counseling

SUMMARY:
The study was done to investigate the differences between workplace exercises and home-based exercises on pain, function, quality of life, and posture (pelvic inclination angle and lumbar lordotic angle) among office workers with non-specific low back pain

DETAILED DESCRIPTION:
Low back pain is the most common musculoskeletal disorder among office workers and a leading cause of disability, affecting psychological well-being and quality of life. Approximately 85% to 95% of cases are categorized as non-specific, with chronic low back pain presenting when symptoms last over 12 weeks. Office workers, who often engage in sedentary tasks, face increased risks of low back pain linked to factors such as physical attributes and psychological stressors like mental fatigue and anxiety. It is suggested that people with low back pain exercise, but there is still debate about whether exercise at work is better than exercise at home. This gap in understanding drives the need for a randomized controlled trial to assess the impact of both interventions on pain, function, quality of life, and posture in office workers with non-specific low back pain

ELIGIBILITY:
Inclusion Criteria:

1. Forty-eight patients with non-specific low back pain of both genders; their ages will range from 25 to 40 years old.
2. Three years of experience at least
3. Eight to ten hours of daily work, at least.
4. Work for 5 days per week.
5. Reported pain intensity from 3 to 7 on a visual analogue scale.
6. Office Workers with body mass index (25 - 29.9 kg/m².
7. Low physical activity levels according to the International Physical Activity Questionnaire (short form).

Exclusion Criteria:

1. Spine pathology.
2. Back surgical operations.
3. Congenital anomalies.
4. Cardiopulmonary and neurological diseases
5. Pregnancy.
6. Postural deformities.
7. Inflammatory diseases.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
assessment of pain intensity | at baseline and after 4 weeks
  The researcher will ask the patient to express how potent he/she feels current pain or the last 24 hours' pain by choosing a point on a 100 mm line drawn between two ends one end refers to the absence of pain and the other refers to the worst intense pain

SECONDARY OUTCOMES:
assessment of activity of daily living | at baseline and after 4 weeks
  The Arabic version of the Modified Oswestry Disability Index is a self-administered questionnaire consisting of ten sections, each with six items that evaluate the limitations in daily living activities. Scores range from 0 to 5, with higher scores indicating greater disability. The final index score is calculated by summing the scores, adjusting for unanswered questions, and expressing it as a percentage. Completion takes approximately 3.5 to 5 minutes, with scoring taking about 1 minute. Scores categorize disability levels: 0%-20% (minimal), 20%-40% (moderate), 40%-60% (severe), 60%-80% (crippled), and 80%-100% (bedbound or exaggerating).
assessment of functional health and well-being | at baseline and after 4 weeks
  The Arabic Version of the 36-Item Short Form Health Survey is a generic tool to measure Quality of Life (QoL) through 36 questions, yielding an 8-scale profile of functional health: Physical Functioning, role limitations due to Physical Problems, Bodily Pain, General Health, Vitality, Social Functioning, role limitations due to emotional problems, and Mental Health. It includes a single-item scale on health transition. The first four subscales form the Physical Composite Scale, and the last four form the Mental Composite Scale, with scores ranging from 0 to 100; higher scores indicate better health and functional status.
assessment of pelvic tilting | at baseline and after 4 weeks
  The Palpation Meter procedure involves subjects standing with feet shoulder-width apart and focusing on a fixed point to minimize posture sway. With arms crossed, an examiner palpates the anterior and posterior superior iliac spines. The caliper tips of the Palpation Meter device are then positioned on these landmarks to measure pelvic inclination, with the procedure repeated three times to calculate an average for statistical analysis.
assessment of lumbar lordotic angle | at baseline and after 4 weeks
  using Baseline Inclinometer. Participants will stand comfortably with arms at their sides while the T12 and S1 spinous processes are marked. The iliac crest serves as a baseline for L4-L5 identification. The investigator will palpate from L4-L5 to S1 and locate T12 using the 12th rib. A bubble inclinometer, zeroed against a bubble level, will be used to measure lumbar lordosis at T12-L1 and S1-S2, with angles recorded and summed.
assessment of physical Activity | at baseline and after 4 weeks
  The Arabic Version of The International Physical Activity Questionnaire (Short-Form) aims to assess physical activity by querying workers about their engagement in various activities over the past week. Respondents will provide details on the type, frequency (in days per week), and duration (in hours and minutes per day) of these activities. The questionnaire evaluates physical activities based on their intensity, classifying them as vigorous (like aerobic walking, running, and jogging), moderate (such as brisk walking, regular home workouts, and leisure swimming), and normal walking, which contributes to the comprehensive assessment of physical activity levels.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Cairo university, Cairo, Egypt